CLINICAL TRIAL: NCT02128516
Title: Controlled, Randomized, Parallel, Double-blind Study of the Effect of NUTRALYS® Pea Protein Supplementation Versus Whey Protein and Placebo on the Muscle Mass and Strength of Volunteers Engaged in Training
Brief Title: NUTRALYS® Pea Protein Oral Supplementation Effects on Muscle Mass
Acronym: nutralys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolas Babault (Other)
Collaborators: Roquette Freres (Industry)
Responsible Party: Sponsor-Investigator, Nicolas Babault, Scientific and sports coordinators, University of Burgundy
Organization: University of Burgundy (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: CEN1118
Record Dates: First submitted 2014-04-24; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
MeSH Terms: interventions — Powders; Whey; Aspartame; Salts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- whey protein (Active Comparator): whey protein
  Interventions: Other: oral powder in sachet
- placebo (Placebo Comparator): placebo
  Interventions: Other: oral powder in sachet
- pea protein (Experimental): pea protein
  Interventions: Other: oral powder in sachet

INTERVENTIONS:
Other: oral powder in sachet
  Other Names: Sachet for oral use composed of proteins (pea or whey) and/or other components (fat-reduced cocoa, flavouring, aspartame, salt, silica dioxide)

SUMMARY:
this clinical trial would try to confirm whether NUTRALYS®, a fast pea protein with an intermediate profile, rich in leucines and other essential amino acids, can significantly enhance muscle mass gain during strength training. This study will compare the efficacy of NUTRALYS® to a reference product. If the results of the study demonstrate a significant improvement in relation to the placebo, not inferior to that of whey, NUTRALYS® could be considered as an alternative to sports nutrition products, to which many people are intolerant.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects from 18 to 35 years of age:
* engaged in moderate or occasional sports activity;
* having given their written informed consent;
* in gainful employment or a student;
* in possession of a medical certificate of fitness for sports

Exclusion Criteria:

* Subject already engaged in regular sports or training increasing muscle strength or volume in the upper limbs and particularly the biceps brachial;
* Subject engaged or having engaged in the last 6 months in weight training more than once a week;
* Subject having had a muscle injury in the 3 months prior to the study;
* Asthmatic subject liable to be administered corticosteroids;
* Subject taking part in another trial;
* Subject with a known hypersensitivity to whey or pea proteins;
* Subject deprived of their freedom for administrative, medical or legal reasons or not in possession of the legal or ethical capacity to enter into a contract due to cognitive function impairment;
* Subject liable not to comply with the constraints required by the protocol;
* Subject not covered by health insurance;
* Subject having taken in the previous month or currently taking: medication, a dietary supplement, sports drink, food for particular nutritional uses or functional foods, of any kind, liable or described as liable to increase physical performance and notably to increase muscle mass;
* Subject taking anabolic protein or corticosteroid treatment;
* Subject on a high-protein diet.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Biceps brachial thickness measured using ultrasonography | 12 weeks after first ingestion
  biceps muscle thickness measured in millimeter using images from ultrasonography

SECONDARY OUTCOMES:
Elbow flexor strength | 12 weeks after first ingestion
  Elbow flexors muscle strength measured in Newton meter using a Biodex isokinetic dynamometer in concentric, eccentric and isometric conditions.
Biceps circumference | 12 weeks after first ingestion
  the circumference of the arm in three sites (proximal, middle and distal) using a tape (centimeter)
body weight | 12 weeks after first ingestion
  Body mass in kg on a scale
tolerance | 12 weeks after first ingestion
  Tolerance measured by quantifying adverse events
muscle force | 12 weeks after first ingestion
  maximal weight lifted during an arm curl exercise (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Francois A Allaert, MD, Principal Investigator — CEN Nutriment
Locations (1):
- Centre d'Expertise de la Performance, Dijon, France

REFERENCES:
- [Derived] Babault N, Paizis C, Deley G, Guerin-Deremaux L, Saniez MH, Lefranc-Millot C, Allaert FA. Pea proteins oral supplementation promotes muscle thickness gains during resistance training: a double-blind, randomized, Placebo-controlled clinical trial vs. Whey protein. J Int Soc Sports Nutr. 2015 Jan 21;12(1):3. doi: 10.1186/s12970-014-0064-5. eCollection 2015. PMID 25628520